CLINICAL TRIAL: NCT03308591
Title: Clinical Efficacy of the Neoadjuvant Chemotherapy for IB2 and IIA2 Stage Cervical Cancer Patients, A Multicenter, Prospective and Randomized Controlled Trial
Brief Title: Clinical Efficacy of the Neoadjuvant Chemotherapy for IB2 and IIA2 Stage Cervical Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, chief physician, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSEM GOG-005B
Record Dates: First submitted 2017-10-08; First posted 2017-10-12 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cervical Neoplasm; Cervical Cancer; Uterine Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NACT (Experimental): The patients will receive 2 courses of platinum based chemotherapy before surgery, 2-3 weeks after each course, doctors will appraise the effect of the chemotherapy. Patients who are sensitive to the treatment will undergo radical hysterectomy and pelvic lymph node dissection 3 weeks after chemotherapy. And 2-3weeks after the surgery, patients will receive adjuvant chemotherapy according to the pathological risk factors.
  Interventions: Drug: NACT; Procedure: RT+PLND; Drug: Adjuvant chemotherapy
- PST (Active Comparator): The patients in this group will undergo radical hysterectomy and pelvic lymph node dissection directly, and 2-6 weeks after the surgery, they will receive adjuvant chemotherapy according to the pathological risk factors.
  Interventions: Procedure: RT+PLND; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: NACT — Platin based chemotherapy
  Arms: NACT
Procedure: RT+PLND — radical hysterectomy+pelvic lymphadenectomy
Drug: Adjuvant chemotherapy — Platin based chemotherapy

SUMMARY:
In recent years, the patients with IB2 and IIA2 stage cervical cancer are still treated with radiotherapy and chemotherapy based treatment, but the radiotherapy will severely damage the function of ovary, cause endocrine dyscrasia and the sexual function of vagina. So we want to study whether neoadjuvant chemotherapy without radiotherapy will achieve the same outcome compared with traditional therapy including radiotherapy. So we randomly divide IB2 and IIA2 stage cervical cancer patients into two groups. The neoadjuvant chemotherapy group will receive two courses of chemotherapy basically composed of platinum, and then undergo surgery, after that, doctors will add more courses of chemotherapy according to the situations of the patients, including whether the patients have the adverse prognostic factors. The control group will undergo surgery directly, and then receive chemotherapy and radiotherapy at the same time. Then we will compare the outcomes of these two groups, and analyze the therapeutic effect, the impact on survival rate and the effect on improving the living quality of patient from two groups. All the outcomes will be fed back to clinical doctors and instruct them to choose better treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis IB2 or IIA2 stage cervical cancer;
* age less than or equal to 65 years old;
* laboratory examination results: WBC ≥ 4*10^9/L, NEU ≥ 20*10^9/L, PLT ≥ 80*10^9/L, serum bilirubin ≤ 2 multiples of the upper normal limit, aminopherase ≤ 2 multiples of the upper normal limit. BUN ≤ normal limit, CR ≤ normal limit;
* KARNOFSKY score ≥ 60;
* No prior treatment;
* pathological diagnosis before surgery is invasive squamous cell carcinoma of cervix;
* well-compliance and willing to keep in touch;
* willing to participate in this study, and sign the informed consent;

Exclusion Criteria:

* participate in other drug clinical trials at the same time;
* respiratory depression, airway obstruction and hypoxia;
* heart diseases (cardiac function at grade II, III or above);
* hematological diseases;
* obvious dysfunction of liver and kidney (above 3 multiples of the upper normal limit);
* a history of brain dysfunction;
* unable to receive surgery and/or unsuitable for radiotherapy or chemotherapy;
* drug abuse or a history of drug abuse;
* unable or unwilling to sign informed consents;
* unable or unwilling to follow the protocols;

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) of the neoadjuvant chemotherapy Group | Up to 3-year
  DFS was definite as the time from randomization to disease recurrence (including death from recurrence if it was the first manifestation of recurrence), death without recurrence.

SECONDARY OUTCOMES:
DSF of the synchro-chemoradiotheraphy group | Up to 3-year

OTHER OUTCOMES:
chemotherapy- and radiotherapy- related adverse effects respectively in two groups | Up to 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The individual participants data will be preserved in the hospital, and all the chemical or physical examination results will be kept in the medical records, the researches, ethics committee and the drug administration will be permitted to look up all the records as we planned. And all the reports or papers about this research will not relate to the patients' identity. But we do not decide whether the information be available to others, the final decision maybe decided by all the patients in this research.

REFERENCES:
- [Derived] Hu Y, Han Y, Shen Y, Chen J, Chen Y, Chen Y, Tang J, Xue M, Hong L, Cheng W, Wang D, Liang Z, Wang Y, Zhang Q, Xing H, Zhang Y, Yi C, Yu Z, Chen Y, Cui M, Ma C, Yang H, Li R, Long P, Zhao Y, Qu P, Tao G, Yang L, Wu S, Liu Z, Yang P, Lv W, Xie X, Ma D, Wang H, Li K. Neoadjuvant chemotherapy for patients with international federation of gynecology and obstetrics stages IB3 and IIA2 cervical cancer: a multicenter prospective trial. BMC Cancer. 2022 Dec 5;22(1):1270. doi: 10.1186/s12885-022-10355-3. PMID 36471257